CLINICAL TRIAL: NCT03543930
Title: Physiologic Effects of CPAP After Vascular Surgery
Acronym: PhyCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Prof., University of Genova
Other Study IDs: PhyCUS Study
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Complications; Respiratory Failure
MeSH Terms: conditions — Postoperative Complications; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major open vascular surgery: Surgical procedures on the abdominal aorta requiring median abdominal incision
  Interventions: Device: Postoperative preventive CPAP
- Endovascular aortic repair: Abdominal aortic repair with endovascular approach
  Interventions: Device: Postoperative preventive CPAP

INTERVENTIONS:
Device: Postoperative preventive CPAP — Administration of a course of 2 hours of CPAP with 7.5 cmH2O pressure and 0.30 FIO2

SUMMARY:
This study aims to investigate, with a case-crossover design, the effects of a short course of preventive CPAP administered in the immediate postoperative period in patients at high-risk of developing postoperative pulmonary complications undergoing major vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Open or endovascular surgery on the abdominal aorta
* Surgical procedure requiring general anaesthesia and invasive intraoperative mechanical ventilation
* Intermediate-high risk of postoperative pulmonary complications (ARISCAT score ≥ 26)

Exclusion Criteria:

* Prolonged post-operative invasive ventilation
* Invasive or non-invasive ventilation or oxygen therapy in the last month
* ASA class IV or V
* Emergency procedures
* Pneumothorax or active pulmonary infection
* Any contraindication to CPAP
* Prolonged bed rest
* Patient refusal to participate or to receive preventive CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing vascular surgical procedures on the abdominal aorta with open or endovascular approach
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-05-25 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
PaO2/FIO2 ratio | Two hours after the administration of CPAP
  Increase of the PaO2/FIO2 ratio compared to the baseline value

SECONDARY OUTCOMES:
Esophageal pressure-time product (PTPes) | Two hours after the administration of CPAP
  Increase of the PTPes compared to the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ball, MD, Principal Investigator — Università degli Studi di Genova
Locations (1):
- Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No